CLINICAL TRIAL: NCT03658408
Title: 4-aminopyridine Treatment for Nerve Injury From Radical Retro-Pubic Prostatectomy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This record should not have been created for this study. It is under another sponsor's account.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ahmed Ghazi, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 72666
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Prostate Disease
MeSH Terms: conditions — Prostatic Diseases | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4-aminopyridine (Experimental): Participants with recent prostatectomies receiving 4-aminopyridine
  Interventions: Drug: 4-aminopyridine
- Placebo (Placebo Comparator): Participants with recent prostatectomies receiving placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 4-aminopyridine — Oral tablet of 2.5 mg given 4 times a day
  Arms: 4-aminopyridine
Drug: placebo — 2.5 mg sugar pill given orally 4 times a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the study drug 4-aminopyridine (4-AP) can help speed up the recovery of peripheral nerve injury after prostatectomy. 4-AP is a potassium channel blocker used to improve walking in multiple sclerosis patients. Investigators will measure the effect that 4-AP may have on the recovery of sexual function and urinary incontinence after prostatectomy.

ELIGIBILITY:
Inclusion Criteria

* Male patients with organ-confined, non-metastatic prostate cancer (stages cT1c-T2c), planning to undergo Robotic-Assisted Laparoscopic Bilateral Nerve sparing radical prostatectomy (NSRP)
* Prostate-specific antigen (PSA) levels less than 10 ng/ml, with biopsy-proven prostate cancer, for whom postoperative adjuvant therapy (e.g. radiation or androgen deprivation therapy) is not expected to be needed
* Ages 45-75
* An International Index of Erectile Function-Erectile Function (IIEF-5) score of greater than or equal to 17 at time of screening
* Is sexually active for at least 6 months with sexual activity within 6 weeks preceding prostate biopsy or surgery.
* Willingness to participate and able to provide informed consent

Exclusion Criteria

* Planned adjuvant therapy after NSRP based on specimen pathology and stage of prostate cancer (stage T3 or greater), positive lymph nodes or positive surgical margins.
* History of prior phosphodiesterase inhibitor use
* Neo-adjuvant therapy prior to NSRP
* History of recurrent prostate cancer
* History of seizures, multiple sclerosis, stroke or any other diagnosed neurological disorder
* History of non-organ confined or metastatic prostate cancer (clinical Stages T3 or greater)
* History of known hypersensitivity to AMPYRA® or 4-aminopyridine
* Patients with history of penile surgery other than circumcision or endoscopic urethral stricture surgery.
* Renal impairment based on calculated GFR (GFR<60 mL/min)
* Use of any other aminopyridine medications for any other indication

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must have prostate disease (only males)
Enrollment: 0 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
percentage of participants with normal erectile dysfunction | 2 months
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.

SECONDARY OUTCOMES:
the time point at which the highest number of subjects reporting normal erectile dysfunction | baseline to month 12
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 3
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 4
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 6
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 8
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 10
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 12
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 14
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 16
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 18
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 20
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 22
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal erectile dysfunction | week 24
  Erectile dysfunction will be assessed using the International Index of Erectile Function. Normal will be defined as a return to baseline. The index ranges from 0-75 with higher scores indicating better outcome. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
percentage of participants with normal urinary continence | 2 months
  Incontinence will be assessed using the Michigan Incontinence Symptom Index. The Michigan Incontinence Symptom Index ranges from 0-40 with higher scores indicating more problems with urinary incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States